CLINICAL TRIAL: NCT02535572
Title: Focal Electrically-Administered Seizure Therapy (FEAST): Studies at Two Enrolling Sites to Further Test and Refine the Treatment
Brief Title: Focal Electrically-Administered Seizure Therapy (FEAST) Studies at Two Enrolling Sites to Further Test and Refine the Treatment
Acronym: FEAST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00042678
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Depression
Keywords: Electroconvulsive Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- FEAST (Experimental): Patients will receive the FEAST form of ECT
  Interventions: Device: FEAST
- RUL UB (Active Comparator): Patients will receive the standard of care, right unilateral ultrabrief ECT (RUL UB)
  Interventions: Device: RUL UB

INTERVENTIONS:
Device: FEAST — FEAST is a new form of ECT, with directional current, rather than traditional alternating current which goes in both directions between the electrodes.
  Arms: FEAST
Device: RUL UB — This is right unilateral ultrabrief ECT, the standard of care.
  Arms: RUL UB

SUMMARY:
This open label investigation further evaluates the safety, efficacy and potential mechanisms of action of a new form of electroconvulsive therapy (ECT). The investigators have recently completed preliminary open-label studies with FEAST, first at Columbia University, and then at the Medical University of South Carolina in Charleston (Nahas et al., 2013b). The investigators have published the outcomes of the first 17 patients studied. One patient withdrew from the study after a single titration session. After the course of FEAST (median 10 sessions), there was a 46.1 + 35.5% improvement in Hamilton Rating Scale for Depression (HRSD24) scores compared to baseline (33.1 + 6.8, 16.8 + 10.9; P < 0.0001). Eight of 16 patients met response criteria (≥50% decrease in HRSD24) and 5/16 met remission criteria (HRSD24≤10). Patients achieved full re-orientation (4 of 5 items correct) in 5.5 + 6.4 min (median time = 3.6 min), timed from when their eyes first opened after treatment. The investigators have now studied 18 more patients (see results below), and we are completing the study in the original IDE with another two more patients still to enroll.

This work allowed us to refine the treatment. For example, the investigators selectively modified the electrode geometry to decrease interelectrode resistance. Additionally the investigators modified the titration schedule, now only administering a standard 800 ma ultrabrief pulse, and thus no longer titrating in the current domain.

In this next proposed trial we will continue to gather efficacy and safety data, and compare these to a parallel non-randomized group receiving ECT standard of care.

ECT is typically delivered in a dynamically adaptive manner, with each person having a different number of treatments, averaging between 8-12 treatment over 4-5 weeks. We thus have to use imprecise time points such as 'at the end of the acute treatment course' rather than specified dates or visits.

DETAILED DESCRIPTION:
This study will provide preliminary evaluation of the following:

1. Further characterization of the efficacy of FEAST and the safety of the treatment.

   1. The primary efficacy measure will be the 24-item Hamilton Rating Scale for Depression. The changes in these scores from before to immediately following the treatment course (typically after 4 weeks) will be compared in patients treated with the FEAST methodology and matched to nonrandomized patients at our facilities who were treated with conventional ECT methods (ultrabrief right unilateral [RUL] ECT).
   2. Acute and subacute cognitive side effects following FEAST will be assessed with a brief neuropsychological battery. The primary acute measures will be the time to return of orientation following seizure induction. The primary subacute measures will be assessment of retrograde amnesia for autobiographical information. The neuropsychological measures will be compared in the patients treated with the FEAST methodology (under this IDE) and matched (but nonrandomized) patients who are treated with conventional ECT methods (also covered under this IDE).
   3. Safety will also be determined by examining the number and frequency of serious adverse advents and adverse events.
2. Characterization of the focal nature of the seizure onset with FEAST and RUL ECT. We will use two main methods to address the issue of focality.

   1. Resting state fMRI before and after a course of FEAST (or conventional RUL ECT). We will address whether FEAST causes changes in hyper connected prefrontal cortical subcortical networks, and whether such an effect is more restricted to prefrontal cortex with FEAST relative to conventional RUL ECT.
   2. Peri-ictal EEG acquired immediately before, during and immediately after the FEAST seizure. We will acquire this in all patients at all treatment sessions. Again, for comparison, we will use identical EEG acquisition methods in patients treated with conventional RUL ECT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Episode
* Pretreatment Hamilton Depression Score >21
* ECT indicated
* Willing and able to give informed consent

Exclusion Criteria:

* History of schizophrenia, schizoaffective disorder, other functional psychosis, or rapid cycling bipolar disorder
* History of central nervous system illness or insult other than conditions associated with psychotropic exposure (e.g., tardive dyskinesia)
* Alcohol or substance abuse or dependence in the past year (DSM-V)
* Secondary diagnosis of a delirium, dementia, or amnestic disorder (DSM-V), pregnancy, or epilepsy
* Requires especially rapid antidepressant response due to suicidality, psychosis, inanition, psychosocial obligations, etc.
* No anticonvulsant mood stabilizers (e.g., Depakote, Tegretol, Lamictal); No lithium; No psychostimulants (e.g., Ritalin, Adderall);

Allowed medications during FEAST/ECT:

Antidepressants, including buproprion Atypical antipsychotics; Hypnotics for sleep; Anxiolytics (limited to up to 3 mg equivalents/day lorazepam)

* ECT in the past six months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-08; Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S George, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Georgia Regents Medical Center, Augusta, Georgia
  - Medical University of South Carolina Brain Stimulation Division, Charleston, South Carolina

REFERENCES:
- [Background] Nahas Z, Short B, Burns C, Archer M, Schmidt M, Prudic J, Nobler MS, Devanand DP, Fitzsimons L, Lisanby SH, Payne N, Perera T, George MS, Sackeim HA. A feasibility study of a new method for electrically producing seizures in man: focal electrically administered seizure therapy [FEAST]. Brain Stimul. 2013 May;6(3):403-8. doi: 10.1016/j.brs.2013.03.004. Epub 2013 Mar 16. PMID 23518262
- [Derived] Youssef NA, George MS, McCall WV, Sahlem GL, Short B, Kerns S, Manett AJ, Fox JB, Dancy M, Cook D, Devries W, Rosenquist PB, Sackeim HA. The Effects of Focal Electrically Administered Seizure Therapy Compared With Ultrabrief Pulse Right Unilateral Electroconvulsive Therapy on Suicidal Ideation: A 2-Site Clinical Trial. J ECT. 2021 Dec 1;37(4):256-262. doi: 10.1097/YCT.0000000000000776. PMID 34015791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 participants were recruited, however only 41 subjects received treatment. 7 subjects withdrew before the treatment began for the following reasons:changed their mind about research (2), time contraints (3), financial reasons (1), no longer met inclusion criteria (1).
Groups:
- RUL UB (Right Unilateral Ultrabrief Electroconvulsive Therapy): Patients will receive the standard of care, right unilateral ultrabrief ECT (RUL UB)
  RUL UB: This is right unilateral ultrabrief ECT, the standard of care.
Period: Overall Study
Arm/Group | FEAST | RUL UB (Right Unilateral Ultrabrief Electroconvulsive Therapy)
Started | 21 | 20
Completed | 17 | 17
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Population: The participants in baseline analysis were those that maintained inclusion criteria throughout the duration of the study. 2 participants were not counted in the baseline analysis population due to exclusionary circumstances.
Groups:
- Total: Total of all reporting groups
Arm/Group | FEAST | RUL UB | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.15 (12.68) | 43.16 (16.44) | 44.17 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Depressive Symptoms as Assessed by Hamilton Rating Scale for Depression
Description: The 24-item Hamilton Rating Scale for Depression has a range score of 0-7 (no depression) 7-17(mild depression) 17-24 (moderate depression) 25 and higher (severe depression). The Hamilton Rating Scale for Depression has a range of 0-72.
  Lower score represents mild depression to no depression at all. A score of 21 or higher for clinical depression (inclusion criteria to participate in study).
Time Frame: From Baseline to end of acute course (typically after 4 weeks)
Measure: Mean (Standard Deviation); unit: percentage of change in score
Arm/Group | FEAST | RUL UB
Number analyzed (Participants) | 20 | 19
percentage of change in score | 60.83 (18.36) | 61.81 (20.80)

2. Primary Outcome: Time to Return to Orientation
Description: Acute and subacute cognitive side effects following FEAST will be assessed with a brief neuropsychological battery. The primary acute measures will be the time to return of orientation following seizure induction. The neuropsychological measures will be compared in the patients treated with the FEAST methodology (under this IDE) and matched (but nonrandomized) patients who are treated with conventional ECT methods (also covered under this IDE).
Time Frame: From Baseline to end of the acute course (typically after 4 weeks)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FEAST | RUL UB
Number analyzed (Participants) | 20 | 19
minutes | 6.56 (5.03) | 8.79 (5.83)

3. Primary Outcome: Retrograde Amnesia for Autobiographical Information Using CUAMI-SF Consistency Scores
Description: Columbia University Autobiographical Memory Interview (CUAMI-SF) assesses the percent consistency in responses and has a maximum of 100%, with lower percentages representing increasing inconsistency. In this interview subjects receive points for each question they answer at Baseline and again at study follow-up, and are graded on the consistency of their answers.
Time Frame: 4 weeks
Population: intent to treat sample
Measure: Mean (Standard Deviation); unit: percentage of consistent responses
Arm/Group | FEAST | RUL UB
Number analyzed (Participants) | 20 | 19
percentage of consistent responses | 69.64 (15.08) | 64.66 (9.83)

4. Secondary Outcome: Number of Adverse Events
Description: Safety will also be determined by examining the number and frequency of serious adverse advents and adverse events from the start of the study through the six month follow up.
Time Frame: From the start of the study through the six month follow up
Population: Participants that met inclusion criteria and are included in the analysis group
Measure: Number; unit: adverse events
Arm/Group | FEAST | RUL UB (Right Unilateral Ultrabrief Electroconvulsive Therapy)
Number analyzed (Participants) | 20 | 19
adverse events
  headache | 108 | 99
  nausea | 35 | 50
  muscle ache | 32 | 46

ADVERSE EVENTS:
Time Frame: Adverse events have been collected throughout the duration of the study, from the beginning of the treatments through the 6 month follow up.
Arm/Group | FEAST | RUL UB
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/19
Other Adverse Events (participants affected / at risk) | 17/20 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FEAST (N=20) | RUL UB (N=19)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Spontaneous Abortion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FEAST (N=20) | RUL UB (N=19)
prolonged seizure (Nervous system disorders) | 1 (1) | 0 (0) — midazolam was required to stop a prolonged seizure in one participant
postictal agitation), (Nervous system disorders) | 1 (1) | 0 (0) — agitation post seizure
postictal delirium (Nervous system disorders) | 0 (0) | 1 (1) — delirium post seizure
headache (Nervous system disorders) | 16 (108) | 17 (99)
Nausea (Gastrointestinal disorders) | 7 (35) | 10 (50)
muscle ache (Musculoskeletal and connective tissue disorders) | 10 (32) | 14 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT02535572/Prot_SAP_000.pdf